CLINICAL TRIAL: NCT03714945
Title: Prospective Longitudinal Study on the Association Between Treatment of Allergic Rhinitis and Cognitive Ability in Children
Brief Title: Study on Association Between Treatment of Allergic Rhinitis and Cognitive Ability in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Michael Tong, Professor and Chairman, Chinese University of Hong Kong
Other Study IDs: CREC Ref No.: 2017.548
Record Dates: First submitted 2018-09-22; First posted 2018-10-22 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Children; Cognitive Ability
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group with Allergic Rhinitis: - Inclusion Criteria
  1. Both genders of 11-14 years, diagnosed with allergic rhinitis on basis of screening instruments, medical history, clinical assessment (by general ORL examination including nasal endoscopy)
  2. Chinese in ethnicity
  3. Positive skin prick test with wheal diameter >= 3mm
  4. Ability to understand the nature, scope, and possible consequences of the study
  5. Capability and willingness to comply with the requirements of the protocol
  Interventions: Other: No intervention
- Control Group without Allergic Rhinitis: - Inclusion Criteria
  1. Both genders of 11-14 years
  2. Chinese in ethnicity
  3. Subjects who have not been diagnosed with a long term medical or psychiatric problem
  4. Subjects who are not currently undergoing any long term medical treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is required as this study is observational.

SUMMARY:
Pilot study on the association between allergic rhinitis and cognitive ability in 174 children aged 11-14 within the same year group at school in which 140 Allergic Rhinitis subjects and 34 non-Allergic Rhinitis subjects. Primary outcome measures include cognitive tests (Trait Making Test, Digit Span Test, Stroop Test, Chinese Auditory Verbal Learning Test, Verbal Fluency Test), so as to assess the cognitive ability of allergic rhinitis patients before and after treatment compared to a control group. Rhinitis Symptom Utility Index (RSUI) of patients will be the secondary outcome measured through questionnaires. Positive skin prick test and endoscopy examination (taking place in Prince of Wales hospital) will be required before the diagnosis of allergic rhinitis. The data will be analysed by the Multilevel models.

DETAILED DESCRIPTION:
INTRODUCTION Allergic rhinitis is the reportedly second most common reported chronic health condition in Hong Kong children under the age of 14, with the Child Health Survey 2005-2006 indicating a prevalence of 24.5%. Allergic rhinitis is a type I hypersensitivity reaction, which occurs when IgE antibodies are produced against allergens, leading to the activation of mast cells which release inflammatory mediators. Common allergens in Hong Kong include house dust mite and cockroaches. Allergic rhinitis causes a multitude of symptoms including itching, sneezing, nasal discharge, post-nasal drip, and nasal congestion. It can cause poor quality sleep, leading to daytime sleepiness, decreased cognitive ability, mood instability and fatigue. Allergic rhinitis leading to a reduction in quality of life in adults has been well established, leading to impediment of cognitive processes and poorer ability in attention-requiring activities (e.g. driving). These symptoms can similarly significantly impede a child's education and quality of life. It is estimated that up to 90% of allergic rhinitis patients are untreated, insufficiently treated, or inappropriately treated.

With regards to children and teenagers, some studies have suggested that allergic rhinitis can cause significant cognitive difficulties, with detrimental effects on children's education and examination performance, however others suggest there is no association. A longitudinal cohort study in 2014 on the treatment of allergic rhinitis in children showed an improvement in attention and divided attention after 1 year of treatment. There are little studies regarding the effect of treatment of allergic rhinitis on cognitive abilities in children.

RESEARCH OBJECTIVES

1. To investigate, if any, the differences between normal and allergic rhinitis patients in terms of cognitive function
2. To investigate the impact of allergic rhinitis on different areas of cognitive function
3. To investigate the improvement of cognitive function in children after 8 weeks of standard treatment of allergic rhinitis

RESEARCH HYPOTHESIS Children with allergic rhinitis are expected to have a heightened improvement in cognitive abilities after the treatment compared to the normal control group due to relief of their nasal symptoms.

STUDY DESIGN This study is a prospective longitudinal pilot study to take place from 15 1 Nov Dec 2017 to 31 Dec 2018. Final report will be completed 30 June 2019.

STUDY SAMPLE AND SETTING The study is to be performed in Hong Kong, with subjects aged 11-14 studying Form 1 and 2 in secondary school being recruited. Recruitment and cognitive testing will take place at the secondary school, whilst physician follow up and skin prick tests will take place at Prince of Wales Hospital. Healthy individuals as well as patients with a history of allergic rhinitis will be recruited. Chinese will be the main language used. The total number of the Form 1 students within the school will be around 200. The estimated participation rate will be approximately 70%. As the prevalence of allergic rhinitis in Hong Kong children under the age of 14 is approximately 24.5%, the expected number of Allergic Rhinitis participants and non-Allergic Rhinitis participants are 140 and 34 respectively.

ELIGIBILITY:
Inclusion Criteria:

- Control Group- Inclusion Criteria

1. Both genders of 11-14 years
2. Chinese in ethnicity
3. Subjects who have not been diagnosed with a long term medical or psychiatric problem
4. Subjects who are not currently undergoing any long term medical treatment.

Patient Group- Inclusion Criteria

1. Both genders of 11-14 years, diagnosed with allergic rhinitis on basis of screening instruments, medical history, clinical assessment (by general ORL examination including nasal endoscopy)
2. Chinese in ethnicity
3. Positive skin prick test with wheal diameter >= 3mm
4. Ability to understand the nature, scope, and possible consequences of the study
5. Capability and willingness to comply with the requirements of the protocol

Exclusion Criteria:

1. Subjects with co-existing nasal conditions other than AR, which may affect nasal pathology (nasal polyposis, sinusitis, severe deviations of nasal septum, tumours of the nasal cavity, acute/chronic rhinosinusitis or any underlying pathology that might affect nasal breathing or nocturnal sleep)
2. Subjects with prior nasal surgery (e.g. nasal cavity, sinuses)
3. Subjects with known brain disorders, prior brain surgery or history of stroke
4. Subjects diagnosed with learning disability, autism or attention deficit hyperactivity disorder (ADHD)
5. Subjects with history of known sleep disorder, central or obstructive sleep apnea, narcolepsy, insomnia, patients requiring regular sleep medication and those hypersensitive to applied topical nasal steroids
6. Subjects who have taken topical nasal steroids, oral anti-histamines or medications affecting nasal symptoms 30 days prior to commencement of study
7. Subjects with hypersensitivity reactions towards topical nasal steroids or oral anti-histamines
8. Subjects previously diagnosed with any psychiatric disorders
9. Subjects who suffered from a respiratory tract infection within the past 30 days
10. Subjects who have clinically major cardiovascular, respiratory, hepatic, neurological, endocrine, immunological or other major systemic disease(s)
11. Subjects who are undergoing a long-term medical treatment plan

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Students aged 11 to 14 currently studying Form 1 and 2 currently studying in secondary schools in Hong Kong will be recruited directly through invitation. Recruitment will include patients suffering from untreated allergic rhinitis in additional to healthy individuals to serve as a control group. Patients suffering from allergic rhinitis will be classified according to ARIA guidelines into mild/moderate/severe, and duration into intermittent/persistent. Patients suffering from rhinitis due to non-allergic origins or those associated with nasal polyposis or sinusitis will be excluded. Patients are going to complete the Rhinitis Symptom Utility Index (RSUI) questionnaire for assessing pre and post symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Trait Making Test (TMT) | 8 weeks
  It tests how fast and accurate the subjects can connect all numbered dots and alphabets in specified instruction. Shorted completion time with accurate compliance to instructions denotes higher score.

SECONDARY OUTCOMES:
Rhinitis Symptom Utility Index (RSUI) | 8 weeks
  Examining the self-reported severity of Rhinitis symptoms. The low score the subject obtained, the more severe level in Allergic Rhinitis symptoms observed.
Stroop Test (Chinese Translated Victoria Version) | 8 weeks
  It tests how fast and accurate subjects call the name of color on alphabet but not the name of the alphabet. Shorter time with accurate identification denotes higher score.
Digit Span Test (DST) | 8 weeks
  It tests the number of correct sequences of a series of digit. Longer sequence of a series of digit denotes higher score.
Chinese Auditory Verbal Learning Test | 8 weeks
  It tests the short-term memory and delayed memory after listening to a series of words in few trials. More words remembered means higher score.
Verbal Fluency Test | 8 weeks
  It tests the verbal fluency of subject who names words in specific topic. More words name within a certain period of time means higher score obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chi Fai CF Tong, MD, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] New Publication by HKU Paediatricians : 'Allergic Rhinitis - The Paediatric Disease You Must Learn' - All News - Media - HKU. (n.d.). Retrieved October 10, 2017, from http://www.hku.hk/press/news_detail_6527.html
- [Background] Aetiology of allergic rhinitis in Hong Kong. (2015, March 19). Retrieved October 10, 2017, from http://www.sciencedirect.com/science/article/pii/S1323893015315343
- [Background] Vuurman EF, Vuurman LL, Lutgens I, Kremer B. Allergic rhinitis is a risk factor for traffic safety. Allergy. 2014 Jul;69(7):906-12. doi: 10.1111/all.12418. Epub 2014 May 9. PMID 24815889
- [Background] Allergic rhinitis: impact, diagnosis, treatment and management. (2016, August 09). Retrieved October 10, 2017, from http://www.pharmaceutical-journal.com/research/review-article/allergic-rhinitis-impact-diagnosis-treatment-and-management/20201509.article
- [Background] Walker S, Khan-Wasti S, Fletcher M, Cullinan P, Harris J, Sheikh A. Seasonal allergic rhinitis is associated with a detrimental effect on examination performance in United Kingdom teenagers: case-control study. J Allergy Clin Immunol. 2007 Aug;120(2):381-7. doi: 10.1016/j.jaci.2007.03.034. Epub 2007 Jun 8. PMID 17560637
- [Background] Jauregui I, Mullol J, Davila I, Ferrer M, Bartra J, del Cuvillo A, Montoro J, Sastre J, Valero A. Allergic rhinitis and school performance. J Investig Allergol Clin Immunol. 2009;19 Suppl 1:32-9. PMID 19476052
- [Background] Kim DK, Rhee CS, Han DH, Won TB, Kim DY, Kim JW. Treatment of allergic rhinitis is associated with improved attention performance in children: the Allergic Rhinitis Cohort Study for Kids (ARCO-Kids). PLoS One. 2014 Oct 17;9(10):e109145. doi: 10.1371/journal.pone.0109145. eCollection 2014. PMID 25330316
- [Background] Lo PS, Tong MC, Revicki DA, Lee CC, Woo JK, Lam HC, van Hasselt CA. Rhinitis Symptom Utility Index (RSUI) in Chinese subjects: a multiattribute patient-preference approach. Qual Life Res. 2006 Jun;15(5):877-87. doi: 10.1007/s11136-005-4828-x. PMID 16721647
- [Background] Lee T, Yuen K, Chan C. Normative data for neuropsychological measures of fluency, attention, and memory measures for Hong Kong Chinese. J Clin Exp Neuropsychol. 2002 Aug;24(5):615-32. doi: 10.1076/jcen.24.5.615.1001. PMID 12187445
- [Background] Hitch JG, McAuley E. Working memory in children with specific arithmetical learning difficulties. Br J Psychol. 1991 Aug;82 ( Pt 3):375-86. doi: 10.1111/j.2044-8295.1991.tb02406.x. PMID 1954527
- [Background] Kremer B, den Hartog HM, Jolles J. Relationship between allergic rhinitis, disturbed cognitive functions and psychological well-being. Clin Exp Allergy. 2002 Sep;32(9):1310-5. doi: 10.1046/j.1365-2745.2002.01483.x. PMID 12220469
- [Background] Den Hartog HM, Derix MM, Van Bemmel AL, Kremer B, Jolles J. Cognitive functioning in young and middle-aged unmedicated out-patients with major depression: testing the effort and cognitive speed hypotheses. Psychol Med. 2003 Nov;33(8):1443-51. doi: 10.1017/s003329170300833x. PMID 14672253
- [Background] Pendleton MG, Heaton RK, Lehman RA, Hulihan D. Diagnostic utility of the Thurstone Word Fluency Test in neuropsychological evaluations. J Clin Neuropsychol. 1982 Dec;4(4):307-17. doi: 10.1080/01688638208401139. PMID 7174838
- [Background] Ardila A, Pineda D, Rosselli M. Correlation between intelligence test scores and executive function measures. Arch Clin Neuropsychol. 2000 Jan;15(1):31-6. PMID 14590565
- [Background] Norrman G, Falth-Magnusson K. Adverse reactions to skin prick testing in children - prevalence and possible risk factors. Pediatr Allergy Immunol. 2009 May;20(3):273-8. doi: 10.1111/j.1399-3038.2008.00761.x. Epub 2009 Feb 10. PMID 19220772
- [Background] International Study of Asthma and Allergies in Childhood Phase II Modules. (1998, May). Retrieved October 10, 2017, from International Study of Asthma and Allergies in Childhood Phase II Modules
- [Background] Downie SR, Andersson M, Rimmer J, Leuppi JD, Xuan W, Akerlund A, Peat JK, Salome CM. Symptoms of persistent allergic rhinitis during a full calendar year in house dust mite-sensitive subjects. Allergy. 2004 Apr;59(4):406-14. doi: 10.1111/j.1398-9995.2003.00420.x. PMID 15005764
- [Background] Adachi, Y., MD, PHD, Yoshida, K., MD, & Itazawa, T., MD. (n.d.). Relationship Between ARIA and ISAAC Questionnaires Regarding to the Classification and Severity of Rhinitis in School Children [Abstract]. Journal of Allergy and Clinical Immunology, 131(2), AB113. Retrieved October 10, 2017, from http://www.jacionline.org/article/S0091-6749(12)03075-8/pdf
- [Background] Goldstein H 1995 Multilevel statistical models. In: Goldstein H, ed. Kendalls library of statistics 3. London: Edward Arnold; 87-94

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03714945/Prot_SAP_000.pdf